CLINICAL TRIAL: NCT03200158
Title: Study on Changes of Barrier and Immune Function in Stress Related Mucosal Disease (SRMD)
Brief Title: Study on Correlated Factors of Barrier and Immune Function in Stress Related Mucosal Disease (SRMD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiuli Zuo (Other)
Collaborators: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor-Investigator, Xiuli Zuo, Deputy director of the physician, Shandong University
Organization: Shandong University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015SDU-QILU-G006
Record Dates: First submitted 2017-05-09; First posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-05

CONDITIONS: Stress Related Mucosal Disease
Keywords: Stress related mucosal disease (SRMD); APACHEII score; C-reactive protein; Malondialdehyde (MDA); transforming growth factor (TGF); interleukin (IL)
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopy biopsy and blood (Other): The healthy volunteers were treated with endoscopy biopsy and blood.The patients were treated with bedside endoscopy biopsy and diagnosed with SRMD due to illness，then collect their blood samples.
  Interventions: Other: Endoscopy biopsy and blood

INTERVENTIONS:
Other: Endoscopy biopsy and blood — Medical operation

SUMMARY:
To study the changes of barrier and immune function in Stress Related Mucosal Disease (SRMD).

DETAILED DESCRIPTION:
38 patients admitted to ICU and 15 healthy volunteers were successively enrolled in this study.The healthy volunteers were treated with endoscopy and biopsy .The 38 patients were treated with bedside gastroscopy and diagnosed with SRMD due to illness. The acute physiology and chronic health evaluation（APACHE）II score were evaluated, malondialdehyde (MDA) as an index of oxygen radical-lipid peroxidation was assessed in the serum. Transforming growth factor(TGF)β1,claudin3, interleukin (IL) 1 and interleukin（IL）10 levels in the gastric mucosa and plasma level of superoxide dismutase(SOD)，Ischemic modified albumin(IMA)and C-reactive protein（CRP）were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Occurrence time: ≤72h.
* With complete clinical data.
* Patients admitted to ICU were treated with bedside endoscopy and diagnosed with SRMD.

Exclusion Criteria:

* Primary digestive tract diseases included stomach cancer, gastric ulcer, cirrhosis with esophagus fundus ventricularis varices and esophageal cancer.
* Patients were complicated with gastric perforation.
* Nonsteroidal anti-inflammatory drugs and antiplatelet agents had been used recently, or with the history of major surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
malondialdehyde (MDA)（nmol/mL） | Month 1
  MDA is an index of oxygen radical-lipid peroxidation was assessed in the serum。Thiobarbituric acid （TBA）method was applied for MDA.
superoxide dismutase(SOD)(u/mL) | Month 1
  The activity of superoxide dismutase(SOD) reflects the the antioxidant ，capacity.Pyrogallol substrate method was applied for SOD.
claudin3 | Month 1
  Tight junctions (TJs) are the most apical component of the intercellular junctional complexes. TJs consist of occludin, the claudin family of proteins, and junctional adhesion molecule (JAM).Among these TJ molecules, claudins are major integral membrane proteins of TJ strands.Studies have shown that H2O2 can change the number of claudin-3.Previously in vitro experiments have reported that H2O2 increases the permeability of the epithelial monolayer by splitting the cell-tight junction complex structure. In our study,the claudin3 in gastric mucosa was measured by western blot method.
TGFβ1 | Month 2
  Measurement of TGFβ1 in gastric mucosa by immunohistochemistry method and microscopic observation.Image-Pro Plus 6.0 software was used to select the same brownish yellow as a uniform standard for determining the positiveness of all photographs. Each photo was analyzed to determine the cumulative cumulative optical density of each photograph.We may collect serm to test TGFβ1 using ELISA method，or we may omit this step.
Acute physiology and chronic health evaluation（APACHE）II score | Month 3
  Acute physiology and chronic health evaluation（APACHE）II score was completed within 24h after admitting, including 12 physiological parameters (each item 0-4 points, total score 0-60 points), age (0-6 points) and chronic disease health status (2-5 points). The total score was 0-71 points. The higher the score, the more severe the illness will be.
interleukin（IL）1β | month 4
  Measurement of interleukin（IL）1β in gastric mucosa by immunohistochemistry method.Image-Pro Plus 6.0 software was used to select the same brownish yellow as a uniform standard for determining the positiveness of all photographs. Each photo was analyzed to determine the cumulative cumulative optical density of each photograph.We may collect serm to test IL1β using ELISA method，or we may omit this step.
interleukin（IL）10 | Month 5
  We measure interleukin（IL）10 in gastric mucosa by immunohistochemistry method.Image-Pro Plus 6.0 software was used to select the same brownish yellow as a uniform standard for determining the positiveness of all photographs. Each photo was analyzed to determine the cumulative cumulative optical density of each photograph.We may collect serm to test IL10 using ELISA method，or we may omit this step.
Nitric oxide synthasei（iNOS） | Month 6
  Measurement of inducible nitric oxide synthasei（iNOS ）in gastric mucosa by immunohistochemistry method.Image-Pro Plus 6.0 software was used to select the same brownish yellow as a uniform standard for determining the positiveness of all photographs. Each photo was analyzed to determine the cumulative cumulative optical density of each photograph.

SECONDARY OUTCOMES:
Ischemic modified albumin（IMA）(u/ml) | Month 7
  Ischemic modified albumin(IMA) is a candidate marker for assessing myocardial ischemia which has been identified as a marker of oxidative stress in a number of studies.Free cobalt colorimetric method was applied for IMA.
C-reactive protein（CRP） | Month 8
  Latex immunoturbidimetric method was applied for C-reactive protein（CRP）.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No